CLINICAL TRIAL: NCT03258684
Title: Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Sepsis and Septic Shock: A Prospective Study
Brief Title: Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Sepsis and Septic Shock
Acronym: HYVCTTSSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Liao Yuping
Record Dates: First submitted 2017-08-15; First posted 2017-08-23 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-01

CONDITIONS: Sepsis
Keywords: corticosteroid; hydrocortisone; septic shock; thiamine; vitamin C
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Hydrocortisone; Ascorbic Acid; Thiamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: The participants in treatment group receive intravenous vitamin C, hydrocortisone, and thiamine. The participants in control group receive normal saline.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin C、hydrocortisone、thiamine (Active Comparator): Intravenous vitamin C (1.5 g every 6 h for 4 days or until ICU discharge), hydrocortisone (50 mg every 6 h for 7 days or until ICU discharge followed by a taper over 3 days), as well as intravenous thiamine (200 mg every 12 h for 4 days or until ICU discharge).
  Interventions: Drug: Hydrocortisone, Vitamin C, and Thiamine
- normal saline (Placebo Comparator): Normal saline 500ml every day for 4 days，then 200ml every day for 3 days.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Hydrocortisone, Vitamin C, and Thiamine — Intervention
  Arms: vitamin C、hydrocortisone、thiamine
Other: Normal saline — Placebo
  Arms: normal saline

SUMMARY:
In this prospective clinical study, the investigators compare the outcome and clinical course of consecutive septic participants treated with intravenous vitamin C, hydrocortisone, and thiamine (treatment group) with a control group treated in the investigators' ICU. The primary outcome is hospital survival. A propensity score is generated to adjust the primary outcome.There is 70 participants in each group.

DETAILED DESCRIPTION:
A prospective randomized controlled trial is conducted.One hundred and forty severe sepsis or septic shock participants admit to the Department of Critical Care Medicine of Zhujiang Hospital,Southern Medical University from September 2017.The participants are divided into control group ( n = 70 ) and treatment group ( n = 70 ).The participants in both groups are treated according to "2016 international guidelines for management of sepsis and septic shock",and the participants in treatment group receive intravenous vitamin C, hydrocortisone, and thiamine. The participants in control group receive normal saline.The patients' clinical and demographic data, including age, sex, admitting diagnosis, comorbidities, requirement for mechanical ventilation, use of vasopressors, daily urine output, fluid balance after 24 and 72 h, length of ICU stay (LOS),and laboratory data (serum creatinine, White Blood Cell (WBC), platelet count, total bilirubin, procalcitonin(PCT), and lactate levels), are recorded.The primary outcome is hospital survival. Secondary outcomes include duration of vasopressor therapy,requirement for renal replacement therapy in patients with Acute kidney injury (AKI), ICU LOS, and the change in serum procalcitonin and Sepsis-Related Organ Failure Assessment (SOFA score) over the first 72 h. Summary statistics are used to describe the clinical data and are presented as means±SD, medians and interquartile range, or percentages as appropriate.Statistical analysis is performed with NCSS 11 (NCSS Statistical Software) and SPSS Statistics version 24 (IBM).

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of sepsis or septic shock (the diagnoses of sepsis and septic shock are based on the 2016 the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3)) and a procalcitonin (PCT) level≥2ng/mL.

Sepsis: Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection.

Septic shock: Septic shock is a subset of sepsis in which underlying circulatory and cellular/metabolic abnormalities are profound enough to substantially increase mortality.

Exclusion Criteria:

* Patients < 18 years of age, pregnant patients, and patients with limitations of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
hospital survival | Up to Day 14

SECONDARY OUTCOMES:
duration of vasopressor therapy | Up to hour 72
requirement for renal replacement therapy in participants with Acute kidney injury(AKI) | Up to Day 14
ICU length of stay(LOS) | Up to Day 14
the change in serum procalcitonin (PCT) | Up to hour 72
Sepsis-Related Organ Failure Assessment(SOFA)score | Up to hour 96

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical Care Medicine of Zhujiang Hospital,Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Derived] Chang P, Liao Y, Guan J, Guo Y, Zhao M, Hu J, Zhou J, Wang H, Cen Z, Tang Y, Liu Z. Combined Treatment With Hydrocortisone, Vitamin C, and Thiamine for Sepsis and Septic Shock: A Randomized Controlled Trial. Chest. 2020 Jul;158(1):174-182. doi: 10.1016/j.chest.2020.02.065. Epub 2020 Mar 31. PMID 32243943
- See also: Related Info — http://dx.doi.org/10.1016/j.chest.2016.11.036